CLINICAL TRIAL: NCT06101446
Title: Evaluation of the Effectiveness of Aromatherapy on Anxiety, Vital Signs, and Postoperative Complications in Lower Impacted Wisdom Tooth Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: YYU-14/20.09.2021
Record Dates: First submitted 2023-09-13; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Tooth, Impacted; Dental Anxiety
Keywords: aromatherapy; lavender oil; wisdom tooth extraction
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lavander Aromatherapy (Experimental): Lavender oil has been known to have calming properties and is one of the most effective aromatherapy oils. It reduces blood pressure and anxiety by stimulating the parasympathetic system.
  Interventions: Other: Lavander Aromatherapy

INTERVENTIONS:
Other: Lavander Aromatherapy — Aromatherapy is one of the potential non-pharmacological methods. Lavender oil has been known to have calming properties and is one of the most effective aromatherapy oils. It reduces blood pressure and anxiety by stimulating the parasympathetic system

SUMMARY:
Dental anxiety is considered to be one of the fears and concerns associated with dental treatment. Lavender has a relaxing and anxiolytic aroma. The aim of this study was to evaluate the effects of aromatherapy on dental anxiety in bilateral impacted wisdom tooth surgery.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral wisdom tooth in mandible

Exclusion Criteria:

* Lavender oil allergy
* Systemic disease
* Off-study drug use
* Smoking
* Pregnancy or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Modified Dental Anxiety Scale (MDAS) | baseline, pre-surgery
  The Modified Dental Anxiety Scale (MDAS) consists of 5 questions each with a 5 category rating scale, ranging from 'not anxious' to 'extremely anxious'. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and MDAS was recorded before each operation.
Modified Dental Anxiety Scale (MDAS) | immediately after the surgery
  The Modified Dental Anxiety Scale (MDAS) consists of 5 questions each with a 5 category rating scale, ranging from 'not anxious' to 'extremely anxious'. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and MDAS was recorded before each operation.
Visual Analog Scale (VAS) Pain Score | 0-7 days
  A Visual Analogue Scale (VAS) is one of the pain rating scales between 1-10. VAS value was recorded (at 3, 6, 12 and 24 hours on day 1 and on days 2, 3, 4, 5, 6 and 7) after each extraction.
Facial Edema | 0-7 days
  Measurement between facial cach extraction.raniometric points (angulus-lateral canthus, tragus-labial commissure, and tragus-pogonion). The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and edema was measured before, 2 days after and 1 week after each operation.
Mouth Opening Measurements | 0-7 days
  Mouth opening measurements is the distance between the incisals of the patient's central teeth at maximal mouth opening.The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and mouth opening was measured before, 2 days after and 1 week after each operation.
Blood Pressure | baseline, pre-surgery
  Blood pressure is the pressure of circulating blood against the walls of blood vessels. Blood pressure was measured with a manual sphygmomanometer.The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and blood pressure was measured before and after each operation.
Blood Pressure | immediately after the surgery
  Blood pressure is the pressure of circulating blood against the walls of blood vessels. Blood pressure was measured with a manual sphygmomanometer.The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and blood pressure was measured before and after each operation.

SECONDARY OUTCOMES:
Oxygen Saturation | baseline, pre-surgery
  Oxygen saturation is a measure of how much hemoglobin is currently bound to oxygen compared to how much hemoglobin remains unbound. Oxygen saturation were measured with a pulse oximeter. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and oxygen saturation was measured before and after operation.
Oxygen Saturation | immediately after the surgery
  Oxygen saturation is a measure of how much hemoglobin is currently bound to oxygen compared to how much hemoglobin remains unbound. Oxygen saturation were measured with a pulse oximeter. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and oxygen saturation was measured before and after operation.
Pulse Rate | baseline, pre-surgery
  The pulse rate is a measurement of the heart rate, or the number of times the heart beats per minute. Pulse rate were measured with a pulse oximeter. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and pulse rate was measured before and after operation.
Pulse Rate | immediately after the surgery
  The pulse rate is a measurement of the heart rate, or the number of times the heart beats per minute. Pulse rate were measured with a pulse oximeter. The number of participants in the split mouth model was 25. A total of 50 impacted teeth were extracted and pulse rate was measured before and after operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl University, Van, Turkey (Türkiye)